CLINICAL TRIAL: NCT03766451
Title: Noninvasive Assessment of Intravascular Volume Status for Postoperative Patients: The Correlation Between Internal Jugular Vein/Common Carotid Artery Cross-Sectional Area Ratio and the Inferior Vena Cava Diameter
Brief Title: Noninvasive Assessment of Intravascular Volume Status for Postoperative Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Hebatullah Negm Eldeen Abd El Azeem, Assistant lecturer, Beni-Suef University
Other Study IDs: Hebatullah Negm Eldeen
Record Dates: First submitted 2018-11-28; First posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Intravascular Volume

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
Ultrasound measurements of the inferior vena cava (IVC) have been proposed as a noninvasive tool to help guide fluid management. Well-established correlations exist between respiratory cycle-induced changes in IVC diameter and C entral Venous Pressure (CVP) . Beyond providing an estimate of CVP, the caval index, or percentage collapsibility of the IVC , has been proposed as a predictor of preload reserve. This noninvasive rapid measurement of CVP is especially important in critical care settings. It can help in differentiating hypovolemic, septic and cardiogenic shock. Changes in volume status will be depicted by change in the diameter of the IVC .

However, the validity and reliability of sonographic assessment of the inferior vena cava have been matters of controversy, and its applicability has been shown to be limited by technical difficulties. Recent study has shown a significant relationship between the internal jugular vein/common carotid artery (IJV/CCA) cross-sectional area ratio and CVP in pediatric burn patients .

DETAILED DESCRIPTION:
Type and Site of The study:

This study will be be done at Beni-Suef university hospital ,Surgical Intensive Care Unit (SICU) after approval of the local ethics and research committee and anesthesia department of Beni- Suef University.

DATE AND PERIOD OF THE STUDY:

The study will be done between NOV. 2018 and Nov. 2019

Patients will be included:

Patients scheduled for elective or emergency major surgeries (e.g., abdominal exploration, cancer bladder, cancer rectum, cancer stomach and aorto-femoral bypass grafting) who require post-operative SICU admission for close monitoring and assessment of volume status will be considered for enrollment.

Thirty five patients will be enrolled in the study; the patients will be admitted to the post-surgical intensive care unit for post-operative close observation and monitoring for at least 24 h. Upon admission, baseline laboratory investigation, chest x-ray, Arterial Blood Gases (ABG) and vital signs (hear rate, mean arterial blood pressure, arterial oxygen saturation and temperature) will be all measured.

Patients will get nurse-controlled analgesia using morphine boluses of 1-2 mg intravenously, followed by a continuous infusion of 1 or 2 mg/h according to the protocol of the SICU team. CVP, sonographic measurement of (IJV/CCA) cross sectional area ratio and IVC diameter will be measured after admitting the patient to SICU as a baseline reading, second measurements will be after achieving CVP between (8-12 cmH2O).

Data to be collected and measured

Demographic data will be obtained from patient's notes and charts including

1- Age, sex, body mass index, ASA physical status and type of surgery.

Cardiorespiratory variables of the Patients include:

* CVP (CMH2O),
* Heart rate (beats/min),
* MAP( mmHg),
* Oxygen saturation (spo2 %),
* Urine output (ml/h),

IVC measurements include:

* IVC Maximum Diameter (cm).
* IVC Minimum Diameter (cm).

Internal jugular vein and common carotid artery measurements include:

* CCA Surface
* IJV surface at inspiration
* IJV surface at expiration
* IJV/CCA RATIO at inspiration
* IJV/CCA RATIO at expiration

Data will be measured after admitting the patient to SICU as a baseline reading, second measurements will be after achieving CVP between (8-12 cmH2O).

ELIGIBILITY:
Inclusion Criteria:.

1. ASA physical status I and II
2. Patients who are able to breathe spontaneously and lay supine post-operative.
3. Patients who had CVP catheter (subclavian or internal jugular vein)

Exclusion Criteria:

* 1- Chronic obstructive or restrictive pulmonary disease. 2-Significant cardiac disease 3-Significant hepatic disease 4-Renal impairment ( creatinine >2 mg/dl). 5- BMI ˃ 30 kg/m2 6- Pneumothorax or mediastinal masses. 7- mechanical ventilation or coming with tracheostomy. 8- defect at the site of sonography. 9- Pregnancy. 10- Instability of vital signs 11- Unwillingness to participate 12- sepsis or septic shock. 13- neurosurgical interventions

Ages: 20 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Patients scheduled for elective or emergency major surgeries (e.g., abdominal exploration, cancer bladder, cancer rectum, cancer stomach and aorto-femoral bypass grafting) who require post-operative SICU admission for close monitoring and assessment of volume status will be considered for enrollment.
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2018-11-10 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
The correlation between (Internal Jugular Vein/Common Carotid Artery Cross-Sectional Area Ratio),and Inferior Vena Cava Diameter by using ultrasound | immediately upon admission to surgical intensive care unit and after acchieving cvp above 8 cmh2o by saline infusion (10 ml/kg) average 3 hours after admission
  The correlation between (Internal Jugular Vein/Common Carotid Artery Cross-Sectional Area Ratio),and Inferior Vena Cava Diameter by using ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Hebatullah Negm eldeen, A.L., Principal Investigator — Beni-Suef University
Locations (1):
- Hebatullah Negm Eldeen, Banī Suwayf, Egypt